CLINICAL TRIAL: NCT04818944
Title: A Pilot, Exploratory Clinical Trial to Evaluate the Safety of Using Continuous IV Infusion of Tirofiban (24 Hours) Including Its Efficacy in Improving Perfusion Post Mechanical Thrombectomy in Acute Ischemic Stroke
Brief Title: Clinical Trial to Evaluate the Safety of Continuous IV Tirofiban in Acute Ischemic Stroke
Acronym: iTREMT
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI has left the Institution
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202010341
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Acute Ischemic Stroke; Ischemic Stroke
Keywords: Mechanical Thrombectomy; Tirofiban; Distal Vessel Reperfusion
MeSH Terms: conditions — Ischemic Stroke | interventions — Tirofiban; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: All study staff is masked to randomization except the following: nursing staff administrating drug, pharmacy staff, statistician, and independent safety assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (tirofiban hydrochloride (AGGRASTAT®)) (Experimental): Subjects will receive an active dose via continuous IV at a rate of 0.10µg/kg/min (actual weight). This rate will begin within one hour of mechanical thrombectomy completion and will be terminated 24 hours after the initial administration time.
  Interventions: Drug: Tirofiban Hydrochloride
- Placebo Arm (Placebo Comparator): Subjects will receive placebo (saline) via continuous IV. This will begin within one hour of mechanical thrombectomy completion and will be terminated 24 hours after the initial administration time.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirofiban Hydrochloride — Tirofiban Hydrochloride will be dosed for 24 hours post MT via continuous IV
  Other Names: Aggrastat
  Arms: Treatment Arm (tirofiban hydrochloride (AGGRASTAT®))
Drug: Placebo — Saline will be dosed for 24 hours post MT via continuous IV
  Other Names: Saline
  Arms: Placebo Arm

SUMMARY:
We will recruit men and non-pregnant women of any ethnic background between the age ≥ 18 and ≤ 90 years that have acute ischemic stroke and underwent Mechanical Thrombectomy (MT) with TICI 2b or 2b following MT. These subject's will be will be randomized to placebo vs. Tirofiban after consent is obtained. This will be administered via continuous IV starting within 60 minutes of MT procedure completion. At the end of the 24 hour continuous IV dosing period a CT angiography and CT perfusion (CTA/CTP) will be obtained. The rest of the subjects inpatient hospital stay will be done per standard of care. The subject's NIHSS and modified Rankin Score (mRS) will be assessed at 90 days.

DETAILED DESCRIPTION:
Procedures:

1. Potential subject present with acute ischemic changes to our Emergency department (ED) and evaluated by stroke neurologist.
2. If the potential subject is a candidate for MT then the patient will be screened for inclusions / exclusions criteria.
3. Patient will undergo MT per standard of care (SOC).
4. At the end of the procedure, the interventionist will assign a specific score for reperfusion following MT.
5. If the interventionist assign a score of TICI 2b, then the potential subject will be eligible to be randomized if she/he meets all the other inclusion /exclusion criteria.
6. If the potential subject has score of TICI 2b after MT and meets all the other inclusion/exclusion criteria, then the power of attorney( POA) /LAR of the potential subject will be approached and informed about the study.
7. If the POA /LAR signs the informed consent, then the subject will be randomized to placebo vs. Tirofiban.
8. The randomization will be 1:1 and will be done by the Investigational Drug Service (IDS) pharmacy.
9. The informed consent must be signed within 60 min from the end of the MT.
10. If the informed consent is obtained, then the agent (placebo or Tirofiban) will must initiated no later than 60 min from the end of the MT.
11. The subject will be transferred to SNICU per SOC.
12. The infusion will continue for 24 hours then stopped.
13. At the end of the 24 hours of infusion a CTA/CTP will be obtained to assess perfusion.
14. If the subject neurological exam deteriorates / worsen during the infusion, the medication will be stopped and unblinded. Non contrast HCT will be obtained immediately to assess if there is a new hemorrhage.
15. If there is hemorrhage and the subject was on Tirofiban then a pack of platelet will be ordered infused immediately. If the subject is on placebo, then no need to infuse a pack of platelets.
16. Platelet count will be assess daily for 48 hours from initiating the medication
17. If the platelet count drops below 20,000, then the medication will be stopped immediately and unblinded.
18. Th rest of the hospitalization will be done per SOC.
19. The subject's NIHSS and mRS will be assessed at 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 90 years
* Acute ischemic stroke (AIS)
* Onset of AIS 6-24 hrs.
* NIHSS score ≥ 6
* AIS due to LVO
* core infarct <30cc or ASPECT score > 6.
* Received MT per SOC
* TICI score of 2B, or TC post MT.
* Able to be imaged by MRI
* Patient or their Legally Authorized Representative (LAR) has provided written informed consent.

Exclusion Criteria:

* Known allergy or hypersensitivity to tirofiban
* Previous stroke in the past 90 days
* Previous intracranial hemorrhage, neoplasm, subarachnoid hemorrhage, or arterial venous malformation
* Clinical presentation suggested a subarachnoid hemorrhage, even if initial CT scan was normal
* Surgery or biopsy of parenchymal organ in the past 30 days
* Trauma with internal injuries or ulcerative wounds in the past 30 days
* Severe head trauma in the past 90 days
* Systolic blood pressure persistently >180mmHg post-MT despite antihypertensive intervention.
* Diastolic blood pressure persistently >105mmHg post-MT despite antihypertensive intervention.
* Serious systemic hemorrhage in the past 30 days.
* Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR >1.5
* Positive urine pregnancy test for women of childbearing potential
* Glucose <50 or >400 mg/dl
* Platelets <100,000/mm3
* Hematocrit <25 %
* Elevated PTT above laboratory upper limit of normal
* Creatinine > 4 mg/dl
* Ongoing renal dialysis, regardless of creatinine
* Received Low Molecular Weight heparins (such as Dalteparin, Enoxaparin, Tinzaparin) in full dose within the previous 24 hours
* Abnormal PTT within 48 hours prior to randomization after receiving heparin or a direct thrombin inhibitor (such as bivalirudin, argatroban, dabigatran or lepirudin)
* Received Factor Xa inhibitors (such as Fondaparinux, apixaban or rivaroxaban) within the past 48 hours
* Received iv tPA
* Pre-existing neurological or psychiatric disease which confounded the neurological or functional evaluations e.g., baseline modified Rankin score >3
* Other serious, advanced, or terminal illness or any other condition that the investigator felt would pose a significant hazard to the patient if tirofiban therapy was initiated a. Example: known cirrhosis or clinically significant hepatic disease
* Current participation in another research drug treatment or interventional device trial
* Informed consent from the patient or the legally authorized representative was not or could not be obtained
* High density lesion consistent with hemorrhage of any degree
* ASPECT score < 6
* Deployment of a stent INTRA and/or EXTRA-cranial
* Did not receive MT
* TICI score of 3 post MT
* Extravasation of contrast during procedure
* Perforation of any vessel during procedure.
* Renal dysfunction
* History of gastrointestinal hemorrhage or major systemic hemorrhage within 30 days, hemoglobin less than 8 g/dL on admission, INR ≥1.5, severe liver impairment as defined as AST, ALT, AP, GGT > 2 x normal
* Creatinine clearance <30 mL/min.
* Major surgery within 30 days with contra-indication to antiplatelet therapy
* Currently pregnant.
* Contraindication for MRI
* Contra-indication to antiplatelet tirofiban:

  1. Active internal bleeding or a history of bleeding diathesis within the previous 30 days
  2. History of thrombocytopenia following prior exposure to AGGRASTAT
  3. History, symptoms, or findings suggestive of aortic dissection
  4. Acute pericarditis
* Actual Body Weight >150kg (due to the lack of safety data)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Intracranial Hemorrhage | Up to 2 weeks post enrollment
  Incidence of intracranial hemorrhage
Infract Size | Up to 2 weeks post enrollment
  Infract size as calculated through imaging methods

SECONDARY OUTCOMES:
Modified Rankin Score | 90 Day post- discharge follow up
  mRS at clinically indicated follow-up visit. Relative frequency of "good outcome" as defined by dichotomized mRS score 0-2
NIH Stroke Scale | 90 Day post- discharge follow up
  NIHSS at clinically indicated follow-up visit.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States